CLINICAL TRIAL: NCT06765473
Title: Comparison Between Preoperative Vaginal and Postoperative Sublingual Misoprostol for Prevention of Postpartum Hemorrhage During Cesarean Section
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Hatem Fouad, resident doctor at Assiut University hospital, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pre-vaginal+ Postperative PPH
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CS group (Active Comparator): women who will undergo elective lower segment CS at term (≥37 weeks) with normal fetal heart tracing
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — preoperative vaginal and postoperative sublingual administration of misoprostol (800 μg) to reducing the amount of blood loss during and 24 hours after CS to determine the optimum time for drug administration.

SUMMARY:
Cesarean section (CS) is one of the most frequently performed operative interventions worldwide [1]. Cesarean section rates increase each year throughout the world. Cesarean delivery can lead to some serious maternal and fetal complications [2] including primary postpartum hemorrhage (PPH). Primary PPH is defined as a blood loss of more than 1000 ml during the first 24 hours after delivery [3], and it is the most common cause of maternal mortality worldwide [4]. Misoprostol is a synthetic prostaglandin E1 analog, commonly used for the prevention and management of PPH. It has potent uterotonic properties and fewer side effects at therapeutic doses [5]; it is absorbed orally, vaginally and across the mucous membranes of the rectum and oral cavity [6] [7] [8]. Misoprostol is affordable, widely available, and easily administrated via multiple routes, and has a good safety profile if properly administrated and monitored, all of which might make it the standard treatment option for PPH in low-resource settings [9]. The benefits (cervical dilatation and uterine contractions) and the adverse effects (nausea, vomiting, diarrhea, fever, and chills) are dose-dependent [10]. Hofmeyr et al. studied the pharmacokinetics of misoprostol administered by various routes. According to this study, the oral route has the most rapid uptake, but the shortest duration. The rectal route has slow uptake but prolonged duration. The buccal and sublingual routes have rapid uptake, prolonged duration and greatest total bioavailability [11]. Besides that, it can be used for termination of pregnancy in cases of missed or incomplete miscarriage [12] [13]. Also, in cases with retained placenta, it may have a role in the management of associated bleeding which mostly results from atony [14] [15]. In the field of gynecology, misoprostol could be used for induction of cervical ripening before office gynecological procedures [16] [17] [18]. This could decrease the associated pain induced by transcervical passage of instruments. Intraoperative blood loss is one of the important complications during CS. In 2011, a systematic review that included twenty-one studies revealed that there is an increased incidence of intraoperative blood loss and blood transfusion with an increased number of cesarean deliveries [19]. Previous reports have shown that misoprostol is effective in reducing blood loss during and after cesarean delivery regardless of route of administration [20] . However, the optimum time for administration of misoprostol to decrease the amount of PPH is still under discussion. A. E. A. Youssef et al. DOI: 10.4236/ojog.2019.94052 531 Open Journal of Obstetrics and Gynecology Therefore the current study aims to compare the effect of preoperative vaginal and postoperative sublingual administration of misoprostol (800 μg) in reducing the amount of blood loss during and 24 hours after CS.

Cesarean section (CS) is one of the most frequently performed operative interventions worldwide [1]. Cesarean section rates increase each year throughout the world. Cesarean delivery can lead to some serious maternal and fetal complications [2] including primary postpartum hemorrhage (PPH). Primary PPH is defined as a blood loss of more than 1000 ml during the first 24 hours after delivery [3], and it is the most common cause of maternal mortality worldwide [4]. Misoprostol is a synthetic prostaglandin E1 analog, commonly used for the prevention and management of PPH. It has potent uterotonic properties and fewer side effects at therapeutic doses [5]; it is absorbed orally, vaginally and across the mucous membranes of the rectum and oral cavity [6] [7] [8]. Misoprostol is affordable, widely available, and easily administrated via multiple routes, and has a good safety profile if properly administrated and monitored, all of which might make it the standard treatment option for PPH in low-resource settings [9]. The benefits (cervical dilatation and uterine contractions) and the adverse effects (nausea, vomiting, diarrhea, fever, and chills) are dose-dependent [10]. Hofmeyr et al. studied the pharmacokinetics of misoprostol administered by various routes. According to this study, the oral route has the most rapid uptake, but the shortest duration. The rectal route has slow uptake but prolonged duration. The buccal and sublingual routes have rapid uptake, prolonged duration and greatest total bioavailability [11]. Besides that, it can be used for termination of pregnancy in cases of missed or incomplete miscarriage [12] [13]. Also, in cases with retained placenta, it may have a role in the management of associated bleeding which mostly results from atony [14] [15]. In the field of gynecology, misoprostol could be used for induction of cervical ripening before office gynecological procedures [16] [17] [18]. This could decrease the associated pain induced by transcervical passage of instruments. Intraoperative blood loss is one of the important complications during

DETAILED DESCRIPTION:
Cesarean section (CS) is one of the most frequently performed operative interventions worldwide [1]. Cesarean section rates increase each year throughout the world. Cesarean delivery can lead to some serious maternal and fetal complications [2] including primary postpartum hemorrhage (PPH). Primary PPH is defined as a blood loss of more than 1000 ml during the first 24 hours after delivery [3], and it is the most common cause of maternal mortality worldwide [4]. Misoprostol is a synthetic prostaglandin E1 analog, commonly used for the prevention and management of PPH. It has potent uterotonic properties and fewer side effects at therapeutic doses [5]; it is absorbed orally, vaginally and across the mucous membranes of the rectum and oral cavity [6] [7] [8]. Misoprostol is affordable, widely available, and easily administrated via multiple routes, and has a good safety profile if properly administrated and monitored, all of which might make it the standard treatment option for PPH in low-resource settings [9]. The benefits (cervical dilatation and uterine contractions) and the adverse effects (nausea, vomiting, diarrhea, fever, and chills) are dose-dependent [10]. Hofmeyr et al. studied the pharmacokinetics of misoprostol administered by various routes. According to this study, the oral route has the most rapid uptake, but the shortest duration. The rectal route has slow uptake but prolonged duration. The buccal and sublingual routes have rapid uptake, prolonged duration and greatest total bioavailability [11]. Besides that, it can be used for termination of pregnancy in cases of missed or incomplete miscarriage [12] [13]. Also, in cases with retained placenta, it may have a role in the management of associated bleeding which mostly results from atony [14] [15]. In the field of gynecology, misoprostol could be used for induction of cervical ripening before office gynecological procedures [16] [17] [18]. This could decrease the associated pain induced by transcervical passage of instruments. Intraoperative blood loss is one of the important complications during CS. In 2011, a systematic review that included twenty-one studies revealed that there is an increased incidence of intraoperative blood loss and blood transfusion with an increased number of cesarean deliveries [19]. Previous reports have shown that misoprostol is effective in reducing blood loss during and after cesarean delivery regardless of route of administration [20] . However, the optimum time for administration of misoprostol to decrease the amount of PPH is still under discussion. A. E. A. Youssef et al. DOI: 10.4236/ojog.2019.94052 531 Open Journal of Obstetrics and Gynecology Therefore the current study aims to compare the effect of preoperative vaginal and postoperative sublingual administration of misoprostol (800 μg) in reducing the amount of blood loss during and 24 hours after CS.

ELIGIBILITY:
Inclusion Criteria:

* The study includes women will undergo elective lower segment CS at term (≥37 weeks) with normal fetal heart tracing

Exclusion Criteria:

* Women with placenta previa . preterm delivery, hypertensive disorders of pregnancy, bleeding tendency, previous history of PPH, concurrent anticoagulant therapy, concurrent long-term use of steroids, fetal distress and antepartum haemorrhage will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
the amount of blood loss | 24 hours
  the amount of blood loss during and 24 hours after CS

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Acharya G, Al-Sammarai MT, Patel N, Al-Habib A, Kiserud T. A randomized, controlled trial comparing effect of oral misoprostol and intravenous syntocinon on intra-operative blood loss during cesarean section. Acta Obstet Gynecol Scand. 2001 Mar;80(3):245-50. doi: 10.1034/j.1600-0412.2001.080003245.x. PMID 11207490